CLINICAL TRIAL: NCT02552589
Title: Clinical Evaluation of the Effect of an Experimental Toothpaste on the Reduction of Dental Plaque and Gingival Inflammation
Brief Title: Effect of Toothpaste on the Reduction of Plaque and Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: Colgate Palmolive (Industry)
Responsible Party: Principal Investigator, Katrin Lorenz, Dr., M.Sc., Assistant Professor, Technische Universität Dresden
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PAR012015
Record Dates: First submitted 2015-09-03; First posted 2015-09-17 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Gingivitis; Dental Plaque
Keywords: clinical trial, phase III; plaque index; gingivitis index; fluoride; toothpaste
MeSH Terms: conditions — Gingivitis; Dental Plaque | interventions — fluorophosphate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test group (Experimental): Amine fluoride toothpaste
  Interventions: Other: Amine fluoride
- Control group (Placebo Comparator): Placebo Sodium monofluorophosphate toothpaste
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Amine fluoride — toothpaste
  Arms: Test group
Other: Placebo — toothpaste
  Other Names: Sodium monofluorophosphate
  Arms: Control group

SUMMARY:
The purpose of this double blind study is to prove whether a fluoride containing toothpaste is able to reduce dental plaque and gingival inflammation in patients who have gingivitis when applied twice daily during brushing at home over a period of 12 weeks.

DETAILED DESCRIPTION:
Before study start, investigators and study nurses will be trained on how to apply SOPs, parameters, and adverse event management. On-site monitoring will be done by the sponsor after recruitment, after visit 2 and after the final visit.

All source data will be entered in paper CRFs. For the statistical analysis these data will be entered into the data bank via double data entry. Programmed range checks, validity checks, consistency checks, and manual/visual data checks for medicinal plausibility will be done before the blind data review meeting. During blind data review meeting minor protocol violations will be recorded and assessed. No imputation of missing data will be done for ITT or PP analyses.

The sample size estimation was carried out by means of one-sided unpaired t-test with a one-sided significance level of α=0.05. For testing superiority of the test product over negative control, the investigators test the hypothesis, H0: μTest product - μNegative control ≤ 0 H1: μTest product - μNegative control > 0 by using a one-sided t-test with α=0.05. A relevant difference of Δ=0.14 and a standard deviation of σ=0.4 was assumed based on previous studies. When estimating a drop-out rate of about 20 % a total of 120 = 102 + 18 subjects per group will be assigned at study start. Drop-outs will not be replaced during the study.

The primary parameter is the difference of plaque index between baseline (V1) value and the value after 12 weeks +/- 5 days (V3) of product use. For primary statistical analysis, a t-tests (unpaired situation) will be performed at a one-sided significance level of α=0.05. The primary efficacy analysis will be performed on the ITT-analysis set.

Secondary variables will be assessed with t-tests and confidence intervals to compare differences between V2, V3, and baseline for test product group and negative control group. Descriptive statistics will be performed for oral examinations for each group (counts and percentages of scores for nominal and ordinal scaled data, for at least ordinal scaled data minimum, maximum, median, mean value and standard deviation).

A two-sided significance level of α=0.05 is chosen for all secondary analyses, no adjustment for multiplicity will be done. Safety assessments will be based mainly on the frequency of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults (aged 18 to 65 years),
* Individuals with gingival inflammation, mean full-mouth GI ≥ 1.2 at inclusion,
* Individuals with plaque, mean full-mouth PI ≥ 1.2 at inclusion,
* Non-smokers or former smokers for at least 1 year or occasional smokers with a maximum of 5 cigarettes per week,
* Individuals who have at least 20 own teeth excluding the wisdom teeth,
* Subjects must have read, understood and signed the informed consent form
* Willingness to abstain from use of interdental brushing devices that contain antibacterial agents, like amine fluoride, chlorhexidine, silver ions etc. during the full course of the study

Exclusion Criteria:

* Individuals who have severe systemic diseases (tumors, infectious diseases) and diseases that require regular systemic medication intake that may affect the gingival condition (e. g. phenytoin, nifedipine, cyclosporine, antibiotics, steroids, antiphlogistics)
* Individuals who have moderate and severe chronic or aggressive periodontitis (PSI > 2 in more than 2 sextants or PSI > 3),
* Individuals who require antibiotic treatments for dental appointments (endocarditis prophylaxis), Individuals treated with antibiotics less than 8 weeks prior to the baseline examination and/or during the duration of the trial,
* Individuals who have participated in another clinical study less than 4 weeks prior to the baseline examination,
* Individuals who have mucosal diseases,
* Individuals who have severe oro-pharyngeal infections,
* Individuals who have significant dental disorders (e.g.: caries, suspected pulp pathology, abscess, pulpitis),
* History of gingival surgery in the previous three month,
* Ongoing dental treatment or any other medical treatment of the oral cavity,
* Individuals who are pregnant or breast feeding,
* Individuals with a history of chronic drug abuse or another illness which does not allow the person to assess the nature and/or possible consequences of the study,
* Smokers with more than 5 cigarettes per week,
* Individuals with known hypersensitivity or allergy to the test products and its ingredients,
* Individuals who were treated with antibacterial mouthrinses (e. g. chlorhexidine) 4 weeks or less before recruitment,
* Individuals unwilling to abstain from additional oral hygiene measures during the treatment phase with exception of their habitual mechanical cleaning procedures,
* Non-Caucasians,
* Subjects can be excluded at the principal investigators discretion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2015-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Plaque index (Silness and Loe 1964) | Change in plaque index from baseline at 12 weeks
  Difference of plaque index, compared between test group and control group.

SECONDARY OUTCOMES:
Plaque index (Silness and Loe 1964) | Change in plaque index from baseline at 3 weeks
  Difference of plaque index, compared between test group and control group.
Plaque index (Silness and Loe 1964) | Change in plaque index from week 3 at 12 weeks
  Difference of plaque index, compared between test group and control group.
Gingival Index (Loe 1967) | Change in gingival index from baseline at 3 weeks
  Difference of gingival index, compared between test group and control group.
Gingival Index (Loe 1967) | Change in gingival index from baseline at 12 weeks
  Difference of gingival index, compared between test group and control group.
Gingival Index (Loe 1967) | Change in gingival index from 3 weeks at week 12
  Difference of gingival index, compared between test group and control group.
Modified Sulcus Bleeding Index (Muhlemann and Son 1971): | Change in bleeding index from baseline at 12 weeks
  Difference of bleeding index, compared between test group and control group.
Modified Sulcus Bleeding Index (Muhlemann and Son 1971): | Change in bleeding index from baseline at week 3
  Difference of bleeding index, compared between test group and control group.
Modified Sulcus Bleeding Index (Muhlemann and Son 1971): | Change in bleeding index from week 3 at week 12
  Difference of bleeding index, compared between test group and control group.
Adverse events | up to 12 weeks from baseline
  List all

CONTACTS AND LOCATIONS:
Locations (1):
- Technische Universität Dresden, Dresden, Germany